CLINICAL TRIAL: NCT04250662
Title: A Randomized, Single Blind, Exploratory Study of the Acute Effects of Guided Imagery and Transcranial Direct Current Stimulation (tDCS) on Electroencephalogram (EEG) Alpha Brain Waves and Pain Levels in Women With Chronic Pelvic Pain
Brief Title: Study of the Acute Effects of Guided Imagery and tDCS on Pain Levels in Women With Chronic Pelvic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled. Lack of patients.
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-362
Record Dates: First submitted 2020-01-27; First posted 2020-01-31 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Pelvic Pain; Chronic Pain
MeSH Terms: conditions — Pelvic Pain; Chronic Pain | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: A single blind, randomized control, exploratory trial to assess the acute effects of tDCS and guided imagery in women with chronic pelvic pain. Qualified individuals will be randomized 1:1:1:1 to receive 1 session of one of the following treatments:
  * 20 minutes of active tDCS with 25 minutes of guided imagery
  * 20 minutes of active tDCS with no guided imagery
  * 20 minutes of sham tDCS with 25 minutes of guided imagery
  * 20 minutes of sham tDCS with no guided imagery
Who Masked: Participant
Masking Description: Device settings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active tDCS with guided imagery (Experimental): Subjects will receive 2 milliamps of electrical stimulation to the brain (transcranial direct stimulation-tDCS) for 20 minutes concurrently while listening to a guided imagery CD specifically designed for women with chronic pelvic pain.
  Interventions: Device: Active tDCS with guided imagery
- Active tDCS alone (no guided imagery) (Experimental): Subjects will receive 2 milliamps of electrical stimulation to the brain (transcranial direct stimulation-tDCS) for 20 minutes while remaining seated, no guided imagery will be provided.
  Interventions: Device: Active tDCS alone (no guided imagery)
- Sham tDCS with guided imagery (Sham Comparator): Subjects will receive 2 milliamps of electrical stimulation to the brain (transcranial direct stimulation-tDCS) for only 30 seconds and then the device will turn off. The device will remain in place, however, for 25 minutes the subject listens to a guided imagery CD specifically designed for women with chronic pelvic pain.
  Interventions: Device: Sham tDCS with guided imagery
- Sham tDCS alone (no guided imagery) (Sham Comparator): Subjects will receive 2 milliamps of electrical stimulation to the brain (transcranial direct stimulation-tDCS) for only 30 seconds and then the device will turn off. The device will remain in place, however, for 25 minutes the subject will remain seated, no guided imagery will be provided.
  Interventions: Device: Sham tDCS alone (no guided imagery)

INTERVENTIONS:
Device: Active tDCS with guided imagery — The subject will be positioned in the sitting/reclining position in a quiet room with the lights dimmed. The tDCS device and audio headphones will be placed on the subject's head. The tDCS device to be used is the Soterix Medical 1X1 device using 2.0 mA of current. The electrodes that will be used will be standard sponge electrodes. The subject will listen to a scripted guided imagery CD specifically developed for women with chronic pelvic pain through the audio headphones. The guided imagery plus active tDCS arm will have 20 minutes of stimulation with 25 minutes of guided imagery.
  Arms: Active tDCS with guided imagery
Device: Active tDCS alone (no guided imagery) — The subject will be positioned in the sitting/reclining position in a quiet room with the lights dimmed. The tDCS device will be placed on the subject's head. The tDCS device to be used is the Soterix Medical 1X1 device using 2.0 mA of current. The electrodes that will be used will be standard sponge electrodes. Active tDCS arm alone without guided imagery, will have 20 minutes of tDCS stimulation without guided imagery.
  Arms: Active tDCS alone (no guided imagery)
Device: Sham tDCS with guided imagery — The subject will be positioned in the sitting/reclining position in a quiet room with the lights dimmed. The tDCS device and audio headphones will be placed on the subject's head. The tDCS device to be used is the Soterix Medical 1X1 device using 2.0 mA of current. The electrodes that will be used will be standard sponge electrodes. The subject will listen to a scripted guided imagery CD specifically developed for women with chronic pelvic pain through the audio headphones. The guided imagery plus sham tDCS arm will have 30 seconds of tDCS stimulation with 25 minutes of guided imagery.
  Arms: Sham tDCS with guided imagery
Device: Sham tDCS alone (no guided imagery) — The subject will be positioned in the sitting/reclining position in a quiet room with the lights dimmed. The tDCS device will be placed on the subject's head. The tDCS device to be used is the Soterix Medical 1X1 device using 2.0 mA of current. The electrodes that will be used will be standard sponge electrodes. Sham tDCS alone arm will have 30 seconds of tDCS stimulation without guided imagery.
  Arms: Sham tDCS alone (no guided imagery)

SUMMARY:
This is a single blind, randomized, exploratory study of transcranial direct stimulation (tDCS) intervention or sham tDCS administered with a standardized guided imagery intervention for chronic pelvic pain. Transcranial Direct Current Sstimulation (tDCS) is a non-invasive brain stimulation therapy. Guided Imagery is a form of hypnosis used to create relaxation.Up to 25 adult women with chronic pelvic pain will be enrolled and randomized (like a flip of a coin). Subjects will remain blinded throughout the study. Subjects will be randomized into one of the following four arms: active tDCS with guided imagery, active tDCS alone (without guided imagery), sham tDCS with guided imagery, or sham tDCS alone (without guided imagery).

DETAILED DESCRIPTION:
Chronic Pelvic Pain (CPP) is a common and often debilitating problem among women. CPP is pain that is felt below the belly button and is severe enough to cause feelings of pressure, pain while sitting or standing for long periods of time, pain with intercourse, painful urination, and pain with bowel movements. Transcranial Direct Current Simulation (tDCS) is a non-invasive brain stimulation technique. As tDCS modulates nerve activity and connectivity, it is also expected to cause measurable changes in brain activity. Guided imagery is a form of hypnosis using words to direct one's thoughts and attention to imagined sensations. Guided imagery has demonstrated efficacy in reducing pain related to many conditions including cancer pain, chronic lower back pain, and post-operative pain. More information is needed to evaluate the effects of tDCS and guided imagery in the treatment of chronic pelvic pain.

The study will consist of one visit. After informed consent is obtained, the following will be collected/completed: health history, demographics, vitals, and questionnaires (BDI, CAGE-AID, PCS, and VAS for pelvic pain). A urinalysis will be collected to assess for infection and a urine pregnancy test for women of child bearing potential. If a subject qualifies they will be randomized. Before treatment, subjects complete an EEG. Treatment will be delivered based on randomization group assignment. After treatment an EEG, VAS, GRA will be collected. Study staff will assess for adverse events during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 to 64 years
* Women must either be unable to become pregnant (surgically sterile or postmenopausal) or must use an approved method of birth control throughout the study period.
* Self-reported CPP defined as pelvic pain that is not related to menstrual cycle and of at lease 6 months duration and refractory to other treatments.
* Subject agrees to not start any new treatments (medication or otherwise) throughout the study participation.
* Subject agrees to maintain stable doses of all current medications throughout study participation.

Exclusion Criteria:

* History of seizures during the last 2 years or diagnosis of epilepsy
* Pacemaker
* Use of carbamazepine, oxcarbazepine, phenytoin, pramipexole or cabergoline within the past 6 months as self-reported
* Parkinson's Disease
* Any condition, including neurological or psychiatric illness, which per investigators' judgment, may increase subject risk
* History of Hunner's lesions
* Lactation, pregnancy, or refusal to use medically approved/reliable birth control in women of child-bearing potential
* Sacral or pudendal Interstim or spinal cord stimulator that is "on"
* Contraindications to tDCS stimulation (e.g. metal in the head, implanted brain medical devices, scalp wounds or infections, etc.)
* History of head injury resulting in more than a momentary loss of consciousness during the last 2 years

Deferral Criteria

1. If a subject has a confirmed UTI, she will be deferred until treatment is completed and symptoms resolve
2. Participating in another intervention study, or received an investigational drug or device within 4 weeks prior to screening
3. Subject received bladder hydrodistention within the past 12 weeks
4. Within the past 4 weeks, initiation of any new medications or any intravesical treatment for treatment of IC/BPS
5. Within the past 24 weeks received any surgery or procedure which may impact the pelvic floor

Note: For the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
To access the acute changes in EEG alpha brain waves in women with CPP after 1 session of each of the following treatments: (1) active tDCS + GI, (2) sham tDCS + GI, (3) sham tDCS alone (no GI) and (4)active tDCS alone (no GI). | Baseline and 48 hours
  An EEG will be collected prior to treatment and after treatment. Changes in alpha waves will be assessed.

SECONDARY OUTCOMES:
To access acute changes in pain in women with CPP after 1 session of each of the following treatments: (1) active tDCS + GI, (2) sham tDCS + GI, (3) sham tDCS alone (no GI) and (4)active tDCS alone (no GI). | Baseline and 48 hours
  Change in pain levels (0-10) on a Visual Analog Scale (VAS) between pre-treatment and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Beaumont Health
Locations (2):
- United States (2):
  - Beaumont Health System, Royal Oak, Michigan
  - Beaumont Hospital-Royal Oak, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No